CLINICAL TRIAL: NCT00583726
Title: Motivational Interviewing for Weight Maintenance
Brief Title: The Women's Healthy Lifestyle Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Zora Djuric, Research Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00012524
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: chemotherapy; exercise; diet; fruit; vegetables; low-fat
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): The control arm receives written information and pedometers
  Interventions: Behavioral: written materials only
- 2 (Experimental): This arm also receives telephone counseling.
  Interventions: Behavioral: motivational interviewing

INTERVENTIONS:
Behavioral: motivational interviewing — telephone counseling
  Arms: 2
Behavioral: written materials only — dietary guidance materials and pedometers
  Arms: 1

SUMMARY:
This study aims to determine if a motivational interviewing counseling style can help women eat a healthy diet and exercise during breast cancer treatment and beyond.

DETAILED DESCRIPTION:
Women receiving chemotherapy for early stage breast cancer often gain weight and body fat, and this contributes to the health burden that cancer survivors face. Weight gain is a concern not only for overall health status, but also as a possible factor for risk of cancer recurrence. Unfortunately achieving weight loss, after a gain has occurred, is difficult, and there are no satisfactory methods for maintenance of weight loss. This study proposes to design and test a novel telephone-based intervention for preventing weight gain during treatment for breast cancer in a pilot, randomized study. The 12-month intervention will target maintenance of current weight and prevention of body fat gain using counseling for moderate exercise and a low-fat, high fruit-vegetable diet. The counseling approach will be based on motivational interviewing techniques and will be delivered through telephone appointments. Motivational interviewing is a client-centered type of counseling that elicits active participation of the patient. By taking a more active role, patients may be more likely to follow through with the recommended lifestyle changes. Study endpoints will include blood markers of dietary compliance, pedometer steps, self-monitoring logs, questionnaires (including quality of life) and anthropometric measures (including body fat by DEXA). An important goal of the study is to establish recruitment methods and demonstrate recruitment rates in newly diagnosed stage I-IIIA breast cancer patients. The study data also will demonstrate implementation of the counseling approach and provide a basis for sample size estimates for a larger trial. This type of intervention, namely a combination of exercise and diet, has been indicated to have good potential for prevention of recurrence. It is therefore necessary to develop effective methods for eliciting these behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Adult female, age 18 and older
* Stage I, II, or IIIA breast cancer
* Scheduled for chemotherapy and completed no more than two weeks of chemotherapy
* Body mass index 25-45 kg/m2
* Stable body weight within 5 pounds in the past 2 months
* Physician approval for participating in a weight control program
* Willing and able to follow advice for exercise and diet quality

Exclusion Criteria:

* Previous invasive cancers, excluding basal cell carcinoma, in the past 10 years
* Following a medically-prescribed diet
* Currently participating in a formal weight loss program
* Medical conditions that preclude safe exercise

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-12; Primary Completion 2010-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in body weight | 12 months

SECONDARY OUTCOMES:
Change in body fat | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zora Djuric, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Djuric Z, Ellsworth JS, Weldon AL, Ren J, Richardson CR, Resnicow K, Newman LA, Hayes DF, Sen A. A Diet and Exercise Intervention during Chemotherapy for Breast Cancer. Open Obes J. 2011;3:87-97. doi: 10.2174/1876823701103010087. PMID 22238561
- [Result] Djuric Z, Ren J, Brown PR, Ellsworth JS, Sen A. Lifestyle factors associated with serum N-3 fatty acid levels in breast cancer patients. Breast. 2012 Aug;21(4):608-11. doi: 10.1016/j.breast.2012.02.003. Epub 2012 Feb 28. PMID 22377591